CLINICAL TRIAL: NCT03146429
Title: Prediction of Future Weight Change With Dopamine Transporter
Status: Completed | Type: Observational
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Kyoungjune Pak, Clinical Assistant Professor, Pusan National University Hospital
Other Study IDs: PusanNUH-2017
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Weight Change, Body
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: I-123 FP-CIT Single photon emission tomography — Brain scan for dopamine transporter

SUMMARY:
This is the re-analyzing study of observational study by Parkinson's Progression Markers Initiative

ELIGIBILITY:
Inclusion Criteria:

* males or females with their age of 30 years or older at screening

Exclusion Criteria:

* subjects with a neurological disorder, a first degree relative with idiopathic PD, Montreal Cognitive Assessment score of 26 or less, medications that might interfere with DAT SPECT scans, anticoagulants that might preclude safe completion of the lumbar puncture, or investigational drugs, and a condition that precludes the safe performance of routine lumbar puncture

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of 192 healthy controls with screening 123I-FP-CIT SPECT.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01-01; Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Weight change | 1, 2, 3, 4, 5 year after SPECT
  weight change per year until 5 years after SPECT